CLINICAL TRIAL: NCT02244086
Title: Analgesic Efficacy of Two Concentrations of Bupivacaine in Women in Labor.
Acronym: EBWL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, María Valeria Jiménez Baez, Investigador Responsable. Coordinador Auxiliar Médico de Investigación en Salud, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: R-2013-2301-21
Record Dates: First submitted 2014-09-03; First posted 2014-09-18 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Obstetric Pain
Keywords: obstetric pain, bupivacaine, analgesic efficacy
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bupivacaine 0.125% (No Intervention): administrate bupivacaine at 0.125% during initiation of effective labor work
- bupivacaine 0.25% (Experimental): Administrate bupivacaine at 0.25% during initiation of effective labor work One of the researchers selected from a randomized list containing pages in both groups with numbers ranging from 0001 to 0110 with 55 pages for each group and these selected folios prepared in sterile form and start the day in the morning, the amount of 10 10 ml syringes with foil for each mixture. The remaining samples were discarded if 10 analgesics are not achieved during the day, and the day new preparations were made.
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: bupivacaine — At the beginning of the work of effective labor maneuver randomly be allocated ( using sealed envelopes) and an outsider to the study prepared the dosage to bupivacaine 0.125% or 0.25% to be administered by epidural catheter for an anesthesiologist to disown the concentration employed. It is measured vital signs, and visual analogue scale dilatation in minutes 0,15,30,60 and 90 after being applied analgesia.
  Other Names: Bupivacaine 0.125%; Bupivacaine 0.25%
  Arms: bupivacaine 0.25%

SUMMARY:
Abstract.

Epidural analgesia is the most safe and effective for the treatment of pain of childbirth method. Epidural Bupivacaine provided excellent analgesia for labor and remains the most widely used local anesthetic in obstetric anesthesia.

Objective: To evaluate the analgesic efficacy of two concentrations of bupivacaine in women in labor.

Methods: 114 patients were included in labor with term pregnancy. Were grouped randomly into two groups: patients who received bupivacaine 0.125 % (Group A) and 0.25% bupivacaine (group B). Patients in group A received 10 ml of 0.125% bupivacaine bolus. The patients in group B received 10 ml. Bupivacaine 0.25% bolus. Pain intensity according to VAS, blood pressure, heart rate, respiratory rate, degree of motor block was assessed using the Bromage scale at different periods of time.

Results: Demographic characteristics and parity were compared, no statistically significant differences. By comparing the values of the VAS measure 0, 15, 30, 60 and 90 minutes into statistically significant differences in favor of the group with 0.25% Bupivacaine with decreased pain perception after 30 minutes, p-value found 0.02. No differences in arterial pressure, heart rate and respiratory rate were found between the two groups.

Conclusion: The concentration of 0.25% Bupivacaine has greater analgesic efficacy compared with 0.125% bupivacaine.

DETAILED DESCRIPTION:
Registration number 2013-2301-21 by Local Committee on Ethics in Health Research and the Mexican Institute of Social Security General Hospital Zone 03. The investigators conduct the study at the Hospital General Regional No. 17 in cancun, Quintana Roo. México. At time in which the obstetrician determined active phase labor and requested obstetric analgesia, patients randomly to one of two study groups being the group A which was administered 0.125% bupivacaine and group B was administered 0.25 % bupivacaine, informed consent for the study was collected.

Blood count, glucose, urea, creatinine and clotting times in the third trimester were included. Preoperative coagulation tests in patients without underlying disease, are expendable if clinical signs of hemorrhage are discarded.

The investigators were masking the patient. The patient was asked for which analgesia bupivacaine unknown concentration that was applied to control the bias of the patient.

Investigators were asking the applicator. One of the researchers selected from a randomized list containing pages in both groups with numbers ranging from 0001 to 0114 with 57 subjects for each group and these numbers selected were prepared in sterile form and start the day in the morning, the amount of 10 ml syringes with foil for each mixture. Ten analgesics were preparing during the day, those not performed bupivacaine were discarded, and the new day preparations were made.

Standardization of the technique and applicator. All anesthesiologists who participated in the study were given a written description of the anesthetic technique used to standardize procedures and avoid bias in the methodology of implementation.

Prior to performing the technique 500 ml of Ringer lactate was infused. Epidural Block (BP) measurement was performed and performed a non-invasive monitoring of heart rate and oxygen saturation monitor electronically. Which were recorded on the data collection sheet designed for this study.

The patient was placed in the left lateral position with knees flexed (fetal position) or sitting. anesthesiologist used surgical clothes, cap and surgical masks, performed surgical handwashing and used sterile gloves and sterile gown and performed surgical toilet of the lumbar back region with iodine solution and sterile drapes were placed delimiting the selected area. Puncture was performed at the level of the L2- L3 with a needle of 17 gauge tuohy -Weiss . Epidural space The search was performed using the technique of loss of resistance to air. The catheter was inserted and left inserted 3-4 cm into the epidural space; was aspirated with a syringe of 3 ml and was determined not to leave blood or cerebrospinal fluid. Sterile prefilled syringe medication to the anesthesiologist who performed the procedure was given; which were injected with either a dose of 10 ml with the corresponding concentration according to the group to which he belonged. Group A or 0.125% bupivacaine dose of 10 ml and group B of 0.25 % bupivacaine. Catheter is firmly fixed to the skin, to prevent their displacement with tape, leaving sealing the proximal end of the epidural catheter. Sensory level as measured by thermal sensitivity this is done with closed eyes of the patient, two test tubes filled, one with cold 5 water use - 10 ° C, and one with hot water at 40-45 ° C, the skin touched the bottom of the tube for more than 3 seconds and was asked to identify the patient saying "cold" or "hot". The region was delimiting with sensory block from zone to zone without blocking lock.

Blocking engine if there was assessed using the modified Bromage scale. which was performed by asking the patient to move his legs or feet and motor block grades were classified as null, partial, complete or almost complete; purposes of numerical comparison gave these categories numbers 0, 1, 2, 3 respectively, where (0) is normal movement of legs and feet (zero ), 1 the patient is able to flex knees with normal movement of feet (part), 2 Unable to flex knees, but with normal foot movement (almost complete ), 3 Unable to move legs or feet (full).

A applied 15 minutes of analgesia again recorded vital signs and note the analgesic level were taken by Visual Analog Scale (VAS), by the responsible investigator which collected the data.

Values Blood Pressure Media (TAM ) < 60mmHg presented the infusion of ringer lactate solution at 5 ml / kg bolus and increase of 5 mg ephedrine was administered iv.

The measurement of the variables involved in the preanalgesia and at 15, 30, 60 and 90 minutes after drug administration were registered.

Variables were measured: Vital signs (blood pressure, heart rate, respiratory rate), sensitive metameric level, engine Block, degree of analgesia according to the VAS.

It was performed according to the following. Metameric sensory level: No blocking, below umbilicus (< T10), between the navel and xiphoid appendix him (T10 - T6), above the xiphoid (> T6). Motor block: 0: can lift both legs straight, 1: You can bend the knee and move your feet, 2: You can only move your feet, 3: You cannot move the lower extremities.

VAS: value between 0 and 10 control / time. 0: no pain 10: Maximum pain imaginable. It was determined by visual analog scale of 0 to 10 cm. Considering effective analgesia according to centimeters decrease from baseline or pre VAS analgesia. Optimal reduction of the initial 4 cm, enough to decrease 3 cm, good with decrease of 2 cm, zero with reduced or unchanged 1cm .

If no analgesic efficacy with VAS valuation at 15 minutes, 5 ml was administered. Mixture used over bupivacaine 0.25% or 0.125 and would restart measurement variables with the set times at 15, 30, 60 and 90 minutes, taking as required for registration and validity of the study variables measuring at least 3 times, if delivery occurs before the scheduled time.

91 minutes was terminated measuring pain analysis records, and records of completion delivery was taken.

Building a database was performed and the statistical program SPSS version 20.0 for Windows 7 was used and proceeded to perform the statistical analysis of data

Analgesic efficacy according to the result of the measurement of the visual analog scale (VAS), according to the result of the evaluation of this scale which is expressed in a numerical value was determined, estimates of frequency measurement were performed, measures dispersion and central tendency for each variable. Comparison of sociodemographic variables (age, number of pregnancy, previous cesarean sections and previous births) and clinical (mild pain, moderate pain, severe pain) that were generated was performed using Student's t test for independent samples, and X2 and trend in the case of nominal variables. To compare differences in variables in blood pressure, heart rate and respiratory rate, EVA, ANOVA for repeated samples was performed.

ELIGIBILITY:
Inclusion Criteria:

* Women with normal pregnancy at term, with active labor, the American Society of Anesthesiologists physical (ASA) st atus I or II.

Exclusion Criteria:

* Patients with problems of language barriers, allergic to local anesthetics, which have been submitted in the last quarter of any of the following situations: pregnancy induced, placenta previa, abnormal fetal variety of presentation, cephalopelvic disproportion, uterine hypertonic hypertensive disease ; Obstetric emergencies such as severe preeclampsia, abruptio placenta detachment, acute fetal distress. Alterations in the anatomy of the spine or previous surgeries that prevent or restrict the conduct of epidural analgesia.

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Decrease in Pain with Visual Analogue Scale (VAS) | 0, 15,30, 60 and 90 minutes
  The visual analogue scale will be measured at the following times: at the time of analgesia, 15 minutes, 30 minutes, 60 minutes and 90 minutes. It will ask the mother after spending the uterine contraction and will show cards that visually validated measure the pain reported by the patient.

SECONDARY OUTCOMES:
cardiac frequency | during labor
  It will be measured with pulse monitor the minute: 0,15,30,60,90 minutes.
Respiratory rate | during labor
  It will be measured with pulse monitor: 0,15,30,60,90 minutes.
Blood pref Blood pressure | during labor
  Be measured with sphygmomanometer calibrated to the minute: 0, 15,30,60 and 90

CONTACTS AND LOCATIONS:
Overall Officials: Maria V Jiménez Báez, PhD, Principal Investigator — Instituto Mexicano del Seguro Social; Ricardo Rodríguez Ramon, Dr., Study Director — Instituto Mexicano del Seguro Social; Ilse C Iparrea Ramos, Dr., Study Chair — Instituto Mexicano del Seguro Social; Horacio Márquez González, MSc, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital General Regional número 17, Instituto Mexicano del Seguro Social., Cancún, Quintana Roo, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rodríguez-Ramón R, Márquez-González H, Jiménez-Báez MV, Iparrea-Ramos IC. Analgesic efficacy of two concentrations of bupivacaine in women in labor: Randomized, controlled, triple blind clinical trial. Colombian Journal of Anesthesiology, Volume 43, Issue 3, July-September 2015, Pages 179-185